CLINICAL TRIAL: NCT00173615
Title: Extracorporeal Membrane Oxygenation Effect in Prolonged Cardiopulmonary Resuscitation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700820
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Cardiopulmonary Resuscitation; Cardiac Arrest; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: ECMO; CPR
MeSH Terms: conditions — Heart Arrest; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Extracorporeal Membrane Oxygenation

INTERVENTIONS:
Procedure: Extracorporeal membrane oxygenation

SUMMARY:
Analysis of the patients' data who were rescued with extracorporeal membrane oxygenation and without ECMO. The survival rate and the weaning rate were analyzed to see the effect of ECMO on the prolonged CPR.

ELIGIBILITY:
Inclusion Criteria:

* CPR > 10 min without return of spontaneous circulation

Exclusion Criteria:

* CPR with traumatic origin unless bleeding was under control, previous irreversible brain damage, terminal status of malignancy, and the age over 75 years. For the patients with post-cardiotomy shock requiring ECLS in the operating theater because of an inability of weaning from cardiopulmonary bypass, they were excluded as well from this ECPR cohort since they did not receive cardiac massage. The patients that had signed "Do-Not-Resuscitate" (DNR) consent were also excluded from ECLS deployment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1996-04; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Sharng Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] KOUWENHOVEN WB, JUDE JR, KNICKERBOCKER GG. Closed-chest cardiac massage. JAMA. 1960 Jul 9;173:1064-7. doi: 10.1001/jama.1960.03020280004002. No abstract available. PMID 14411374
- [Background] Eisenberg MS, Mengert TJ. Cardiac resuscitation. N Engl J Med. 2001 Apr 26;344(17):1304-13. doi: 10.1056/NEJM200104263441707. No abstract available. PMID 11320390
- [Background] Bedell SE, Delbanco TL, Cook EF, Epstein FH. Survival after cardiopulmonary resuscitation in the hospital. N Engl J Med. 1983 Sep 8;309(10):569-76. doi: 10.1056/NEJM198309083091001. PMID 6877286
- [Background] Cooper S, Janghorbani M, Cooper G. A decade of in-hospital resuscitation: outcomes and prediction of survival? Resuscitation. 2006 Feb;68(2):231-7. doi: 10.1016/j.resuscitation.2005.06.012. Epub 2005 Dec 1. PMID 16325314
- [Background] Weil MH, Fries M. In-hospital cardiac arrest. Crit Care Med. 2005 Dec;33(12):2825-30. doi: 10.1097/01.ccm.0000191265.20007.9d. PMID 16352966
- [Background] Chen YS, Chao A, Yu HY, Ko WJ, Wu IH, Chen RJ, Huang SC, Lin FY, Wang SS. Analysis and results of prolonged resuscitation in cardiac arrest patients rescued by extracorporeal membrane oxygenation. J Am Coll Cardiol. 2003 Jan 15;41(2):197-203. doi: 10.1016/s0735-1097(02)02716-x. PMID 12535808
- [Background] Cummins RO, Chamberlain D, Hazinski MF, Nadkarni V, Kloeck W, Kramer E, Becker L, Robertson C, Koster R, Zaritsky A, Bossaert L, Ornato JP, Callanan V, Allen M, Steen P, Connolly B, Sanders A, Idris A, Cobbe S. Recommended guidelines for reviewing, reporting, and conducting research on in-hospital resuscitation: the in-hospital 'Utstein style'. American Heart Association. Circulation. 1997 Apr 15;95(8):2213-39. doi: 10.1161/01.cir.95.8.2213. No abstract available. PMID 9133537
- [Background] Tunstall-Pedoe H, Bailey L, Chamberlain DA, Marsden AK, Ward ME, Zideman DA. Survey of 3765 cardiopulmonary resuscitations in British hospitals (the BRESUS Study): methods and overall results. BMJ. 1992 May 23;304(6838):1347-51. doi: 10.1136/bmj.304.6838.1347. PMID 1611332
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Derived] Chen YS, Lin JW, Yu HY, Ko WJ, Jerng JS, Chang WT, Chen WJ, Huang SC, Chi NH, Wang CH, Chen LC, Tsai PR, Wang SS, Hwang JJ, Lin FY. Cardiopulmonary resuscitation with assisted extracorporeal life-support versus conventional cardiopulmonary resuscitation in adults with in-hospital cardiac arrest: an observational study and propensity analysis. Lancet. 2008 Aug 16;372(9638):554-61. doi: 10.1016/S0140-6736(08)60958-7. Epub 2008 Jul 4. PMID 18603291